CLINICAL TRIAL: NCT05264987
Title: Evaluation of Outcomes of Obstetric Patients With COVID-19 Disease Followed up in the Intensive Care Unit
Brief Title: Outcomes of Obstetric Patients With COVID-19 Disease in the ICU
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Karasu, MD, Principal Investigator, Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 2011-KAEK-25 2021/06-20
Record Dates: First submitted 2022-02-24; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Obstetric Anesthesia Problems; Intensive Care Unit; Morality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: intensive care follow-up — The need for the mechanical ventilator, the length of stay in the intensive care unit, and outcomes of mothers were recorded. Deceased patients were evaluated in detail.

SUMMARY:
Although several studies are conducted in the general population researching the clinical and laboratory parameters predicting the progression to severe disease in COVID-19, the data are very few in obstetric patients. Therefore,the investigators aimed to evaluate the characteristics, prognosis, laboratory parameters, and mortality of obstetric patients followed up in the intensive care unit (ICU) due to severe COVID-19 disease and to determine the factors affecting mortality.

DETAILED DESCRIPTION:
This study was a single-center, retrospective, and observational trial and carried out with the principles of the Declaration of Helsinki. All patient demographics and information were analyzed retrospectively from the patient files.

Demographic data, obstetric histories, comorbidities, treatments received in the intensive care unit (ICU), delivery types, anesthesia types, and outcomes of newborns and mothers were retrospectively evaluated from the medical records. The need for the mechanical ventilator, the length of stay in the ICU, and outcomes of mothers were recorded. Laboratory findings were noted on the first day of admission to the ICU, including routine complete blood count, liver and kidney function, coagulation parameters, C-reactive protein (CRP), and albumin levels. Then neutrophil to lymphocyte (N/L) ratio, platelet to lymphocyte (P/L) ratio, and CRP to albumin (CRP/Alb) ratio were calculated. Deceased patients were evaluated in detail.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients (during the pregnancy and postpartum period, from the beginning of pregnancy and up to 42 days after delivery) hospitalized in the intensive care unit of our tertiary care hospital
* Patients who had positive PCR nasopharyngeal swabs for COVID-19

Exclusion Criteria:

* Patients who had negative PCR nasopharyngeal swabs for COVID-19 and were clinically suspicious

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — obstetric patients
Study Population: Obstetric patients (during the pregnancy and postpartum period, from the beginning of pregnancy and up to 42 days after delivery) hospitalized in the intensive care unit of our tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
intensive care follow-up | up to 200 days
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Derya Karasu, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided